CLINICAL TRIAL: NCT01449123
Title: An Open-label Single Site Single Dose Pilot Study Using Mannitol Challenge Test With the Purpose to Explore Treatment With Fixed Dose Combinations in Adult Subjects With Asthma in Primary Care in Sweden
Brief Title: Mannitol Challenge Test in Adult Asthma Patients With Fixed Dose Combinations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mundipharma AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLT4501; 2011-000939-86 (EudraCT Number)
Record Dates: First submitted 2011-09-08; First posted 2011-10-10 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Asthma
Keywords: Asthma; mannitol challenge test; Sweden; primary care
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inhaler (Experimental): Subjects prescribed fixed dose combinations perform Mannitol Challenge Test and Reversibility Test once
  Interventions: Drug: Mannitol challenge test & reversibility test

INTERVENTIONS:
Drug: Mannitol challenge test & reversibility test — Patients perform an asthma control test (ACT) to establish if they are "well controlled" or "symptomatic". All patients will perform then perform the mannitol challenge test. Aridol™ is an indirect osmotic bronchial challenge test which can be used to identify bronchial hyperresponsiveness

SUMMARY:
The primary objective in this pilot study is to explore if asthma patients prescribed fixed dose combinations (budenosid/formoterol (Symbicort®), salmeterol/fluticasone (Seretide®), beclometasone/formoterol (Innovair®) are optimal treated regarding the mannitol challenge test and the following reversibility test.

The primary endpoint is to identify asthma patients responding positive or negative to the mannitol challenge test and/or the reversibility test.

The hypothesis is that not all patients are well treated.

ELIGIBILITY:
Inclusion criteria

1. Males and females, age 18-65 years.
2. Subjects diagnosed with asthma.
3. Subjects with a baseline FEV1 of ≥70% of the predicted value.
4. Outpatients at primary clinic.
5. Subjects treated with a fixed dose combination for at least the last three months.
6. Subjects who have withheld their asthma- and allergy medication according to individual instructions at the day of the challenge test.
7. Subjects who are able to read and comprehend Swedish and are willing to sign an informed consent.

Exclusion Criteria

1. Subjects with evidence of any other respiratory and/or obstructive disease including recent infection/exacerbation.
2. Subjects treated with a oral corticosteroid within 4 weeks (28 days) prior to the day of the challenge test.
3. Any history of hypersensitivity to mannitol challenge test.
4. Any contraindications to use of the diagnostic study medication.
5. Subjects who are unsuitable for other reason(s) in the opinion of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2011-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Mannitol challenge test (Aridol™) + short-acting β2-agonist - positive response. | One day only (Day 1). Subjects complete an ACT, the mannitol challenge test and the reversibility test. This is the end of the study, there is no follow up.
  For the Primary efficacy variable, positive response Mannitol challenge test (Aridol™) followed by short-acting β2-agonist will be given as number and percentage for the ITT-population, as defined by the following: ≥15% fall in FEV1 from baseline; 10% incremental fall in FEV1 between two consecutive doses in the test; Reversibility test with a short-acting β2-agonist - increase in FEV1 of ≥15% from the last dose of mannitol in the challenge test.

CONTACTS AND LOCATIONS:
Locations (1):
- Näsets Läkargrupp i Höllviken, Höllviken, Sweden